CLINICAL TRIAL: NCT01043081
Title: Prevalence Rates of Sexually Transmitted Infections and Sexual Risk Behaviors Among African American Women Who Have Sex With Women
Brief Title: Sexually Transmitted Infections Among African American Women Who Have Sex With Women
Acronym: WSW
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi State Department of Health (Other Government); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Leandro A. Mena, Associate Professor of Medicine, University of Mississippi Medical Center
Other Study IDs: 2008-0143
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Sexually Transmitted Infections; HIV Infections
Keywords: African American women who have sex with women; Sexually transmitted infections; Homosexuality; Human papillomavirus; Cervical intraepithelial neoplasia; Herpes simplex virus types 1 and 2; Chlamydia; Gonorrhea; Trichomoniasis; Bacterial vaginosis; Syphilis; Human immunodeficiency virus
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections; Homosexuality; Uterine Cervical Dysplasia; Chlamydia Infections; Gonorrhea; Trichomonas Infections; Vaginosis, Bacterial; Syphilis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endocervical and vaginal secretion specimens are being retained for future research studies in this field of sexually transmitted diseases.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the rates of sexually transmitted infections (STI) among a group of African American women who have sex with women (AA WSW). The first study hypothesis is that AA WSW are at risk for acquiring and transmitting STI, including the human immunodeficiency virus (HIV). The second study hypothesis is that AA WSW participate in multiple high-risk sexual activities that may facilitate transmission of STIs, including HIV.

DETAILED DESCRIPTION:
Historically, women who have sex with women (WSW) have been thought to be at low risk for acquiring sexually transmitted infections (STI), presumably due to the absence of genital mucosal contact present during vaginal-penile sex or due to the assumption that the vaginal mucosa experiences a lesser degree of trauma during female sex than during heterosexual sex. This assumption has been challenged and debated over the past two decades. In addition, the sexual health risks of WSW are only beginning to be understood.

To date the majority of research regarding STI in women has occurred in heterosexuals. National and local surveillance data that estimate the risk for STI transmission between WSW are limited, especially among African Americans. This is a group of women that may exhibit distinctive behavioral characteristics that may put them at higher risk for sexually transmitted infections STI and HIV than their Caucasian counterparts. This group of women has traditionally been reluctant to discuss their sexual orientation with physicians for fear of being stigmatized. The burden of STIs, including HIV, experienced by this group of women is largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* African American race
* Sexual contact with another female within the past 6 months
* Ability to give written informed consent

Exclusion Criteria:

* Male
* Age less than 18 years old
* Race other than African American
* No sexual contact with another woman within the past 6 months
* Pregnant
* Prior enrollment in this study
* Participants who, for any reason, in the opinion of the investigator, do not have the ability to give written informed consent or may not be expected to comply with the requirements of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is African American women, aged 18 or above, who present to the Crossroads Clinic (STD Clinic) in the Jackson, MS metropolitan area for STI screening/evaluation who have engaged in sexual contact with another woman within the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence rates of sexually transmitted infections | 18 Months

SECONDARY OUTCOMES:
Associated sexual risk behaviors | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Leandro A Mena, MD, MPH, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Crossroads Clinic, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with investigators

REFERENCES:
- [Result] Muzny CA, Sunesara IR, Griswold ME, Kumar R, Lefkowitz EJ, Mena LA, Schwebke JR, Martin DH, Swiatlo E. Association between BVAB1 and high Nugent scores among women with bacterial vaginosis. Diagn Microbiol Infect Dis. 2014 Dec;80(4):321-3. doi: 10.1016/j.diagmicrobio.2014.09.008. Epub 2014 Sep 16. PMID 25262105
- [Result] Muzny CA, Rivers CA, Parker CJ, Mena LA, Austin EL, Schwebke JR. Lack of evidence for sexual transmission of genital Candida species among women who have sex with women: a mixed methods study. Sex Transm Infect. 2014 Mar;90(2):165-70. doi: 10.1136/sextrans-2013-051361. Epub 2014 Jan 15. PMID 24431188
- [Result] Muzny CA, Sunesara IR, Kumar R, Mena LA, Griswold ME, Martin DH, Lefkowitz EJ, Schwebke JR, Swiatlo E. Characterization of the vaginal microbiota among sexual risk behavior groups of women with bacterial vaginosis. PLoS One. 2013 Nov 13;8(11):e80254. doi: 10.1371/journal.pone.0080254. eCollection 2013. PMID 24236175
- [Result] Muzny CA, Sunesara IR, Austin EL, Mena LA, Schwebke JR. Bacterial vaginosis among African American women who have sex with women. Sex Transm Dis. 2013 Sep;40(9):751-5. doi: 10.1097/OLQ.0000000000000004. PMID 23949590
- [Result] Muzny CA, Sunesara IR, Martin DH, Mena LA. Sexually transmitted infections and risk behaviors among African American women who have sex with women: does sex with men make a difference? Sex Transm Dis. 2011 Dec;38(12):1118-25. doi: 10.1097/OLQ.0b013e31822e6179. PMID 22082722